CLINICAL TRIAL: NCT03377179
Title: A Phase 2 Study of ABC294640 Alone and in Combination With Hydroxychloroquine Sulfate in the Treatment of Patients With Advanced, Unresectable Intra-hepatic, Perihilar and Extra-Hepatic Cholangiocarcinoma
Brief Title: A Study of ABC294640 Alone and in Combination With HCQ Sulfate in the Treatment of Advanced Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-108
Expanded Access: NCT03414489 (No longer available)
Record Dates: First submitted 2017-12-01; First posted 2017-12-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma; Cholangiocarcinoma Non-resectable; Cholangiocarcinoma, Perihilar; Cholangiocarcinoma, Extrahepatic; Cholangiocarcinoma, Intrahepatic
Keywords: Clinical Trial, Phase II; Multicenter Trials; Clinical Study; Clinical Trials, Non-Randomized; Oral capsule; Single arm; Anti-cancer; Anti-inflammatory; ABC294640; Yeliva ®; opaganib; Hydroxychloroquine Sulfate; HCQ; Autophagy
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Part 1- single-arm Phase IIA study, all participants receiving ABC294640, continuously administered in 28 day cycles, until disease progression, unacceptable toxicity or voluntary withdrawal Enrollment in a two-stage design: 12 participants will be accrued, if none of those patients respond, registration will halt. If one or more patients respond, additional 27 patients evaluable for efficacy will be enrolled.
  Part 2- identical to Part 1 with the exceptions: co-treatment of both ABC294640 and HCQ and study will consist of two phases: Phase I, a hybrid accelerate dose escalation run-in starting at HCQ dose of 200 mg QD. Based on safety results, patient cohorts will be expanded and dosing will escalate up to 600 mg BID. Phase II, treatment with ABC294640 and HCQ at the Phase I determined dose. Up to 15 participants evaluable for safety and tolerability will be accrued in Phase I and 20 participants evaluable for efficacy in Phase II, Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABC294640 +/- HCQ treatment (Experimental): Part 1: All participants will be receiving ABC294640, 500 mg twice a day (BID), continuously in 28 day cycles Part 2: All participants will be receiving ABC294640, 500 mg twice a day (BID) and HCQ at a determined level, continuously in 28 day cycles
  Interventions: Drug: ABC294640; Drug: Hydroxychloroquine Sulfate 200 MG

INTERVENTIONS:
Drug: ABC294640 — Two 250 mg capsules of ABC294640 will be taken twice daily
  Other Names: yeliva; opaganib
Drug: Hydroxychloroquine Sulfate 200 MG — HCQ tablets will be taken at a dose that will be determined
  Other Names: HCQ

SUMMARY:
ABC-108 is a single-arm Phase IIA clinical study of ABC294640 (Yeliva ®, opaganib) alone and in combination with hydroxychloroquine sulfate (HCQ) in the treatment of cholangiocarcinoma (CCA). In Part 1 of this clinical study, all participants will be receiving ABC294640 and in Part 2 all participants will be receiving ABC294640 and HCQ to explore the drugs activity signal in CCA. The study drug, ABC294640 is an orally available inhibitor of the enzyme sphingosine kinase-2 (SK2). SK2 is an innovative target for anti-cancer therapy because of its critical role in sphingolipid metabolism, which is known to regulate tumor cell death and proliferation. ABC294640 also inhibits proliferation and induces apoptosis of cholangiocarcinoma cell lines. Furthermore, in a recent Phase I trial, ABC294640 demonstrated clinical activity in CCA patients. HCQ, is an orally available, FDA approved therapy for the treatment of malaria as well as discoid and systemic lupus erythematosus and rheumatoid arthritis. It is also known as an inhibitor of autophagy, a pro-survival mechanism utilized by many cancers. Evidence indicates that inhibition of autophagy can increase the therapeutic activity of ABC294640 in CCA. In Part 1 of this study, ABC294640 will be continuously administrated orally, twice a day, in 28 day cycles. In Part 2, ABC294640 and HCQ will be continuously administrated orally (the safe and tolerable will be determined in the study) in 28 day cycles. Administration of drug/s in both parts of the study will continue until disease progression, unacceptable toxicity or voluntary withdrawal initiated by the participants or physician.

DETAILED DESCRIPTION:
This is an open-label clinical study to explore the activity signal of ABC294640 and of ABC294640 and HCQ in adult subjects who have been diagnosed with unresectable cholangiocarcinoma either intra- perhilar or extra-hepatic. The study will be conducted at 5 sites in the USA.

For Part 1, a maximum of 39 participants evaluable for efficacy will be enrolled in the study. Eligible participants will receive ABC294640, 500 mg twice a day, continuously administered in 28 day cycles.

Part 2 will be a single-arm Phase IIA study identical to Part 1 but treatment will consist of both ABC294640 together with HCQ. Additionally, Part 2, will consist of two phases: Phase I: accelerate HCQ dose-escalation run-in starting with a HCQ dose of 200 mg QD (once a day). Based on safety results, patient cohorts will be expanded, and dosing will continue to 200 mg BID (twice a day), 400 mg BID and 600 BID. At the end of Part2, Phase I, it will be determined what is the safe and tolerable HCQ dose for Phase II.

For Part 2, up to 15 patients evaluable for safety and tolerability will be enrolled in Phase I component of Part 2; and 20 patients evaluable for efficacy in the Phase II component of Part 2. All eligible participants will receive ABC294640, 500 mg BID in addition to the determined HCQ dose, continuously administered in 28 day cycles.

In addition to physical, neurological and eye exams (eye exams only for participants receiving HCQ), blood and urine samples will be routinely collected for safety and to determine response to the study drugs. Participants will be radiographically assessed for disease status every 2 cycles of treatment.

Tumor biopsies, when accessible, will be obtained within 21 days prior to the beginning of treatment and again on the beginning of the second treatment cycle.

All participants will be followed every 2 months for progression and survival for a maximum of 24 months after the last patient has been entered to the study. Follow up procedures may include physical examination, laboratory work and radiographic tumor assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed intrahepatic, perihilar or extra-hepatic CCA.
2. Patients with no more than 2 prior treatments with systemic anti-neoplastic therapy for CCA.
3. The tumor is unresectable and not amenable to curative therapy.
4. One or more tumors measurable on CT scan per RECIST 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0- 1.
6. Life expectancy of at least 3 months.
7. Age ≥18 years.
8. Signed, written IRB-approved informed consent.
9. A negative pregnancy test (if female).
10. Acceptable liver and renal function:

    * Bilirubin ≤ 1.5 times upper limit of normal (CTCAE Grade 2 baseline)
    * AST (SGOT), ALT (SGPT) ≤ 2.5 x upper limit of normal (ULN),
    * Serum creatinine ≤ 1.5 X ULN (CTCAE Grade 1 baseline)
    * Albumin > 3.0 g/dL
11. Acceptable hematologic status:

    * Absolute neutrophil count ≥1000 cells/mm3
    * Platelet count ≥75,000 (plt/mm3) (CTCAE Grade 1 baseline)
    * Hemoglobin ≥ 9 g/dL
12. Acceptable blood sugar control:

    - Fasting glucose value ≤ 160 mg/dL (CTCAE Grade 1 baseline)
13. Urinalysis: No clinically significant abnormalities.
14. Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 X ULN after correction of nutritional deficiencies that may have contributed to prolonged PT/PTT.
15. For men and women of child-producing potential, willingness to use effective contraceptive methods during the study. If female (or female partner of male patient), was either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing one of the following medically acceptable methods of birth control and agreed to continue with the regimen throughout the duration of the study:

    * Oral, implantable or injectable contraceptives for 3 consecutive months before the baseline/randomization visit.
    * Total abstinence from sexual intercourse (≥ 1 complete menstrual cycle before the baseline/randomization visit).
    * Intrauterine device.
    * Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream

Exclusion Criteria:

1. >2 previous systemic anti-neoplastic regimens for CCA.
2. Previously having received ABC294640 or HCQ (or chloroquine) for the treatment of a malignancy.
3. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
4. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
5. Pregnant or nursing women. NOTE: If a woman became pregnant or suspects she is pregnant while participating in this study, she must inform her treating physician immediately.
6. Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 28 days prior to study entry.

   Patients who had received any antineoplastic therapy > 28 days prior to starting treatment with ABC294640 and HCQ must have recovered from the reversible effects of prior antineoplastic therapy (with the exception of alopecia and Grade 1 neuropathy).
7. Unwillingness or inability to comply with procedures required in this protocol.
8. Known infection with human immunodeficiency virus.
9. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
10. Patients who were currently receiving any other investigational agent.
11. Patients who were receiving drugs that were sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes that could not have been stopped at least 7 days or 5 half-lives (whichever was longer) before starting treatment with ABC294640, could not have been replaced with another appropriate medication or not given for the duration of the clinical study must be discussed with the Medical Monitor in order to determine eligibility for the study.
12. Patients who are taking warfarin, apixaban, argatroban or rivaroxaban.
13. If the patient is to receive HCQ, pre-existing retinopathy.
14. Known history of G-6-PD Deficiency, porphyria or psoriasis.
15. History of macular degeneration, visual field changes, retinal disease, or cataracts that would interfere with funduscopic eye examinations.
16. History of allergic reactions attributed to compounds of similar chemical or biologic composition to HCQ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Part1 - Determine Response Rate | At least 4 months
  To determine the response rate (RR) of CCA defined as objective responses (OR), i.e. complete and partial responses (CR, PR) plus stable disease (SD) of at least 4 months to treatment with ABC294640.
Part 2 - Determine the Durable Disease Control Rate | At least 4 months
  To determine the Durable Disease Control Rate (DDCR) of CCA defined as Disease Control Rate (DCR) of at least 4 months duration to treatment with ABC294640 and HCQ

SECONDARY OUTCOMES:
Physical exam to include eye exams (the latter only for patients enrolled in Part 2) to measure safety and tolerability of ABC294640 alone and in combination with HCQ | From screening phase, during beginning of each cycle of treatment, till 30 days after the end of treatment (an estimated median of 5 months)
  A physical exam which will include weight measurment in kilograms will be performed in screening and on the beginning of each cycle of treatment till 30 day post treatment.
A general neurological exam to measure safety and tolerability of ABC294640 alone and in combination with HCQ | From screening phase, during beginning of each cycle of treatment, till 30 days after the end of treatment (an estimated median of 5 months)
  A general neurological exam will be performed in screening and on the beginning of each cycle of treatment till 30 day post treatment.
HADS score for depression and anxiety to measure safety and tolerability of ABC294640 alone and in combination with HCQ | From screening, during each cycle of treatment, till the end of treatment (an estimated median of 4 months). Patient diaries will be filled on a daily basis during treatment.
  HADS (Hospital Anxiety and Depression Scale) questionnaire will be utilized to monitor any alterations in the participant's anxiety and depression levels.
ECOG performance score to measure safety and tolerability of ABC294640 alone and in combination with HCQ | From screening, during each cycle of treatment, till the end of treatment (an estimated median of 4 months). Patient diaries will be filled on a daily basis during treatment.
  ECOG (Eastern Cooperative Oncology Group) performance score to the participant's performance status and how it is impacting the daily living abilities.
MMSE score to measure safety and tolerability of ABC294640 alone and in combination with HCQ | From screening, during each cycle of treatment, till the end of treatment (an estimated median of 4 months). Patient diaries will be filled on a daily basis during treatment.
  MMSE (Mini-Mental State Examination) questionnaire will be utilized for evaluating the mental state of the participants.
Daily diary entries to aid in asessing safety and tolerability of ABC294640 alone and in combination with HCQ | From screening, during each cycle of treatment, till the end of treatment (an estimated median of 4 months). Patient diaries will be filled on a daily basis during treatment.
  Participants will be asked to fill a daily diary to record the drug administration and any side effects that they may experience.
Number of treatment-related Adverse Events alone and in combination with HCQ | From screening till the 30 days after the end of treatment (an estimated median of 5 months)
  Adverse events will be graded according to the revised NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE version 4.03) to measure the safety and tolerability of treatment with ABC294640 alone and in combination with HCQ in patients with unresectable CCA.
The Maximum Plasma Concentration (Cmax) of ABC294640 and of HCQ | From the first day of treatment until the beginning of second cycle of treatment (on day 1, 15, 28 approximately)
  To determine the pharmacokinetics of ABC294640 (Part 1) and of ABC294640 and HCQ (Part 2) in the first 12 patients by measuring Maximum Plasma Concentration (Cmax) of ABC294640 and HCQ
The Area Under the Curve (AUC) of ABC294640 (Part 1) and of ABC294640 and HCQ (Part 2) | From the first day of treatment until the beginning of second cycle of treatment (on day 1, 15, 28 approximately)
  To determine the pharmacokinetics of ABC294640 (Part 1) and of ABC294640 and HCQ (Part 2) in the first 12 patients by measuring the Area Under the Curve (AUC) of ABC294640 and of HCQ which reflects the body exposure to drug after administration of a dose of the drug.
Determine the progression free survival (PFS) | Every 2 months for a maximum of 24 months after the last participant has been entered to the study
Determine Disease Control Rate (DCR=CR+PR+SD) | Every 2 months for a maximum of 24 months after the last participant has been entered to the study
  Determine Disease Control Rate (DCR) = complete response (CR)+ partial response (PR) + stable disease (SD)
Determine the overall survival (OS) | Every 2 months for a maximum of 24 months after the last participant has been entered to the study

OTHER OUTCOMES:
Determine the effect of treatment with ABC294640 alone or in combination with HCQ on pharmacodynamic markers that are associated with the mechanism of action of the drug. | Within 21 days prior to treatment and on the beginning of the second cycle of treatment (approximately a month)
  Tumor biopsies, when accessible, will be obtained and will be assessed for tumor signaling proteins (c-Myc, pAKT, SK2). Peripheral Blood Mononuclear Cells (PBMC) for c-Myc will be collected within 1 hour prior to the pre- and posttreatment biopsies (or at the scheduled time of biopsy if not performed).
Serial measurement of circulating tumor DNA (ctDNA) | Prior to treatment till the end of study (assessed at screening, beginning of cycle three of treatment and every 8 weeks thereafter, up to 24 months)
  Serum ctDNA be assessed for mutational status and development of new mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Borad, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Emory University, Atlanta, Georgia
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding X, Chaiteerakij R, Moser CD, Shaleh H, Boakye J, Chen G, Ndzengue A, Li Y, Zhou Y, Huang S, Sinicrope FA, Zou X, Thomas MB, Smith CD, Roberts LR. Antitumor effect of the novel sphingosine kinase 2 inhibitor ABC294640 is enhanced by inhibition of autophagy and by sorafenib in human cholangiocarcinoma cells. Oncotarget. 2016 Apr 12;7(15):20080-92. doi: 10.18632/oncotarget.7914. PMID 26956050
- [Background] Beljanski V, Knaak C, Smith CD. A novel sphingosine kinase inhibitor induces autophagy in tumor cells. J Pharmacol Exp Ther. 2010 May;333(2):454-64. doi: 10.1124/jpet.109.163337. Epub 2010 Feb 23. PMID 20179157
- [Background] French KJ, Zhuang Y, Maines LW, Gao P, Wang W, Beljanski V, Upson JJ, Green CL, Keller SN, Smith CD. Pharmacology and antitumor activity of ABC294640, a selective inhibitor of sphingosine kinase-2. J Pharmacol Exp Ther. 2010 Apr;333(1):129-39. doi: 10.1124/jpet.109.163444. Epub 2010 Jan 8. PMID 20061445
- [Result] Britten CD, Garrett-Mayer E, Chin SH, Shirai K, Ogretmen B, Bentz TA, Brisendine A, Anderton K, Cusack SL, Maines LW, Zhuang Y, Smith CD, Thomas MB. A Phase I Study of ABC294640, a First-in-Class Sphingosine Kinase-2 Inhibitor, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2017 Aug 15;23(16):4642-4650. doi: 10.1158/1078-0432.CCR-16-2363. Epub 2017 Apr 18. PMID 28420720